CLINICAL TRIAL: NCT06804837
Title: Implement and Test Visual Consent Template and Process
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 202501068; R01HS029310 (AHRQ)
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Alzheimer Disease
Keywords: Informed consent; Key information; Common Rule; Research ethics
MeSH Terms: conditions — Neoplasms; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge randomized control trial to implement and test the consent template and process in three studies. Randomization will occur at the research coordinator/research team level. Each participating research team member will begin in the standard consent arm of the study. Subsequently, they will be randomized to the visual key information page arm at staggered time points to undergo training and begin using the visual key information page with patients who are eligible for the selected research study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Research Staff: Standard Consent (Active Comparator): Each participating research team member will begin in the standard consent arm of the study. The standard consent consists of a summary using text only.
  Interventions: Other: Standard consent
- Research Staff: Visual Consent (Experimental): After beginning in the standard consent arm, the research staff will then be randomized to the visual key information page arm at staggered time points to undergo training and begin using the visual key information page with patients who are eligible for the selected research study. Research staff will also complete a baseline survey to assess feasibility, acceptability, and appropriateness of using visual consent pages as well as their institution's willingness and ability to implement using visual key information pages into routine care. Research staff will also complete a post-study survey on attitudes toward consent, the intervention (feasibility, acceptability, appropriateness of the intervention), organizational readiness for participant engagement, and willingness to continue the invention.
  Interventions: Other: Visual consent
- Participants: Visual Consent (Experimental): Participants will view the visual consent summary and will complete surveys with measures of knowledge, satisfaction with the information, decisional conflict, and potential covariates (i.e., demographics and health literacy).
  Interventions: Other: Visual consent
- Participants: Standard Consent (Active Comparator): Participants will view the standard consent consisting of summary text only and will complete surveys with measures of knowledge, satisfaction with the information, decisional conflict, and potential covariates (i.e., demographics and health literacy).
  Interventions: Other: Standard consent

INTERVENTIONS:
Other: Visual consent — Visual key information page
  Arms: Participants: Visual Consent; Research Staff: Visual Consent
Other: Standard consent — Summary text only
  Arms: Participants: Standard Consent; Research Staff: Standard Consent

SUMMARY:
The investigators plan to conduct a stepped wedge randomized control trial to implement and test the consent template and process in three studies. Randomization will occur at the research coordinator/research team level. Each participating research team member will begin in the standard consent arm of the study. Subsequently, they will be randomized to the visual key information page arm at staggered time points to undergo training and begin using the visual key information page with patients who are eligible for the selected research study.

ELIGIBILITY:
Eligibility Criteria for Patients:

* Adult participants (18+) eligible for one of three participating trials at Washington University, University of Utah, or University of North Carolina at Chapel Hill. The eligibility criteria for the main trials are below:

  * UNC:

    * Basal-like PDAC Treated with Gemcitabine, Erlotinib, and Nab-paclitaxel (PANGEA) trial inclusion criteria:

      * Written informed consent was obtained to participate in the study and HIPAA authorization for release of personal health information.
      * Participant is willing and able to comply with study procedures based on the judgment of the investigator.
      * Age ≥ 18 years at the time of consent.
      * Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
      * Consent to a mandatory pre-study biopsy if archival tissue is not available or sufficient.
      * Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen.
  * Washington University:

    * Returning Research Results That Indicate Risk of Alzheimer Disease Dementia to Healthy Participants in Longitudinal Studies (WeSHARE)

      * Participants of the Knight Alzheimer Disease Research Center.
      * Participants with available results from an Alzheimer Disease blood biomarker test.
      * Participants who agreed to be contacted for additional research studies.
  * University of Utah:

    * Huntsman Cancer Institute Total Cancer Care

      * Participants who have been diagnosed with any type of tumor or cancer.
      * Participants with genetic predispositions or family history of cancer or tumors.
      * Participant volunteers willing to share samples and data for research.

Eligibility Criteria for Research Staff:

* Research staff/coordinators of one of the three participating trials at Washington University, University of Utah, or University of North Carolina at Chapel Hill.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 515 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in feasibility (FIM) of implementation (Research Staff only) | From baseline to end of study (estimated to be 4 months)
  4 items on a Likert scale ranging from completely disagree to completely agree. Higher scores indicate greater feasibility. (1=completely disagree, 3= neither agree nor disagree, 5= completely agree)
Change in acceptability (AIM) of implementation measures (Research Staff only) | From baseline to end of study (estimated to be 4 months)
  4 items on a Likert scale ranging from completely disagree to completely agree. Higher scores indicate greater acceptability. (1=completely disagree, 3= neither agree nor disagree, 5= completely agree)
Change in appropriateness (IAM) of implementation measure (Research Staff only) | From baseline to end of study (estimated to be 4 months)
  4 items on a Likert scale ranging from completely disagree to completely agree. Higher scores indicate greater appropriateness. (1=completely disagree, 3= neither agree nor disagree, 5= completely agree)
Change in organizational willingness and ability to implement strategies (Research staff only) | From baseline to end of study (estimated to be 4 months)
  Measure of organizational readiness for engagement (MORE) measure; 4-point scale (1=not willing, 4=; willing) report mean and SD; higher scores indicate higher level of readiness

SECONDARY OUTCOMES:
Knowledge of information provided in the consent (Participant only) | At time of consent review (day 1)
  The investigators will ask up to7 true/false/unsure questions. Missing responses will be considered false/incorrect. An overall knowledge score will be calculated with the percentage of items correctly answered. Higher scores indicate greater participant understanding of the clinical trial.
Satisfaction of information provided in the consent (Participant only) | At time of consent review (day 1)
  NIH Health Information National Trends Survey (HINTS); 5-items on a Likert scale (1=completely disagree, 3= neither agree nor disagree, 5= completely agree). Higher scores indicate higher satisfaction.
Decisional conflict (Participant only) | At time of consent review (day 1)
  SURE measure; 4-item measure. Scores less than equal to 3 indicate the presence of decisional conflict
Number of enrollments to clinical trials (Participant only) | At time of consent review (day 1)
  The investigators will document whether or not participants enroll in the trials.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - University of Utah Huntsman Cancer Institute (HCI), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Prior to sharing, data will be redacted to strip all identifiers and strategies will be adopted to minimize risks of unauthorized disclosure of personal identifiers. Publicly available documentation will include the survey questions (including any relevant skip patterns), a codebook, univariate statistics for each variable, and study-level metadata. The codebook will include a brief description of each variable along with the question number and question text, variable name, variable label, value labels, and standard codes for missing values-including codes for non-applicable, "don't know," or prefer not to answer.
  User information will be required to access data files. As part of the registration process, users must agree to the conditions of use governing access to the data, including restrictions around redistributing data, destruction of the data after analyses, immediate reporting of any disclosures, and proper acknowledgment of the data resource.
Supporting Information: Study Protocol, SAP
Time Frame: Final submission and release of the study data will occur 12 months following the end of data collection. Study data deposited will be available to the research community in perpetuity. Datasets underlying methodological publications will be shared at or prior to initial publication date.
Access Criteria: Researchers who provide a methodologically sound plan.

REFERENCES:
- [Derived] Cooksey KE, Goldstein EC, Lee CN, Mozersky J, Kaphingst KA, Liu J, Wu S, Volkmar M, Catalan-Gallegos V, Politi MC. Implementing and evaluating visual key information pages compared to text-based key information: protocol for a stepped-wedge cluster randomized trial. BMC Med Ethics. 2025 Nov 29;27(1):1. doi: 10.1186/s12910-025-01341-y. PMID 41318540
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu
- See also: Huntsman Cancer Institute at University of Utah — https://healthcare.utah.edu/huntsmancancerinstitute/
- See also: Lineberger Comprehensive Cancer Center — https://unclineberger.org/